CLINICAL TRIAL: NCT05650229
Title: An Interventional, Randomised, Double-blind, Parallel-group, Placebo-controlled, Flexible-dose, Adaptive Study of the Efficacy of KL1333 in Adult Patients With Primary Mitochondrial Disease
Brief Title: Efficacy of KL1333 in Adult Patients With Primary Mitochondrial Disease
Acronym: FALCON
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abliva AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KL1333 2020-104A
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Primary Mitochondrial Disease
Keywords: Chronic fatigue; Myopathy; Muscle weakness; Exercise intolerance; Diabetes
MeSH Terms: conditions — Muscular Diseases; Muscle Weakness; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- KL1333 (Experimental): Twice daily
  Interventions: Drug: KL1333
- Matching Placebo (Placebo Comparator): Twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KL1333 — Twice daily
  Arms: KL1333
Drug: Placebo — Twice daily
  Arms: Matching Placebo

SUMMARY:
The primary objective of the FALCON study is to evaluate the efficacy of KL1333 on selected disease manifestations of primary mitochondrial disease (PMD) following 48 weeks of treatment. This objective involves evaluating the efficacy of KL1333 versus placebo on fatigue symptoms and impacts on daily living as well as on functional lower extremity strength and endurance. Additionally, the study evaluates the safety and tolerability of KL1333.

DETAILED DESCRIPTION:
The FALCON study is investigating whether the study medicine, KL1333, improves fatigue levels and physical abilities of people living with mitochondrial disease. The investigators are also evaluating the tolerability of the study medicine. For this study, the effects of KL1333 are compared with those from a placebo (a pill that looks like the study medicine but contains no active medicine). The study medicine (or placebo) is a tablet that is taken twice daily during the treatment period of 48 weeks.

Participation in the FALCON study is divided into 3 parts:

* Screening and baseline: 8-12 weeks
* Treatment: 48 weeks
* Safety follow-up: 5 weeks Total duration: 61 - 65 weeks

Patients who complete the screening phase and are enrolled in the study are randomly assigned to receive either the study medicine (KL1333) or placebo (no active medication). Patients are more likely to receive the study medication than placebo (for every five people who take part, three receive KL1333 and two receive placebo). Neither the participants nor the study team know who is receiving the study medicine or placebo and participants are not able to change which treatment they are assigned.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* A confirmed PMD diagnosis caused by a known pathogenic gene mutation or deletion of the mitochondrial genome (category 6 of the International Classification of Inborn Metabolic Disorders [ICIMD])12 according to American College of Medical Genetics (ACMG)/Association of Molecular Pathology (AMP) criteria1, with multisystemic disease expressions, including:

  1. m.3243A>G associated MELAS-MIDD spectrum disorders,
  2. single large scale mtDNA deletion associated KSS-CPEO spectrum disorders,
  3. other multisystemic mtDNA-related disease (including MERRF).
* Presence of chronic mitochondrial fatigue:

  * History of mitochondrial fatigue for at least 3 months prior to the Screening Visit AND
  * Presence of at least moderate level of fatigue, assessed by PROMIS® Fatigue PMD Short form raw score ≥ 27 at Screening and Baseline
* Presence of mitochondrial myopathy defined as:

  * Myopathy (proximal muscle weakness), NMDAS Section III Clinical Assessment, item 5 score ≥ 1, which reads: "minimal reduction in hip flexion and/or shoulder abduction only (e.g. MRC 4+/5)". For the inclusion only hip flexion, but not shoulder abduction, should be taken into account. AND / OR
  * Exercise Tolerance: NMDAS Section I, item 9 score ≥ 1, which reads: "unlimited on flat - symptomatic on inclines or stairs".
* Patients must be able to perform at least 2 repetitions and the maximal capacity must not exceed 17 repetitions in males or 16 repetitions in females in a 30s STS test at screening.
* Clinically stable, apart from symptoms associated with the diagnosis of mitochondrial disease, at Screening and Baseline, as determined by medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations at Screening, as assessed by the investigator.
* The patient is willing and able to attend study appointments within the specified time windows.
* Willingness and ability to complete electronic PROs.
* Willingness to maintain a stable diet during the Screening and study periods.
* Patients who take any mitochondrial disease-focused vitamins or supplemental therapies, including coenzyme Q10 (CoQ10), niacin/nicotinamide (vitamin B3), and L-arginine, has been on a stable dose regimen of these for 3 months prior to randomisation and intends to stay on a stable dose for the duration of the study period.
* Willingness to suspend treatment with idebenone during the study.
* Female patient is not pregnant and at least one of the following conditions apply:

  1. Not a woman of childbearing potential (WOCBP)
  2. WOCBP must agree not to try and become pregnant and use a highly effective method of contraception from the time of informed consent through at least 36 days (~5 half-lives of KL1333 plus 30 days) after the last dose of investigational medicinal product (IMP) administration.
* Male patients with female partner(s) of childbearing potential must agree to use a male condom in addition to using highly effective contraception throughout the treatment period and for 96 days after the last dose of IMP administration. The requirement to use a male condom also applies to male patients with a pregnant or breastfeeding partner.
* Female patients must agree not to breastfeed starting at Screening and throughout the study period and for 36 days after the last dose of IMP administration.
* Female patients must agree to not donate ova throughout the study period and for 36 days after the last dose of IMP administration, and male patients must agree to not donate sperm throughout the study period and for 96 days after the last dose of IMP administration.

Exclusion Criteria:

* Primary mitochondrial disease with predominant neurodegenerative phenotypes, such as, but not limited to, Leigh syndrome, Leber hereditary optic neuropathy (LHON) and Neuropathy ataxia-retinitis pigmentosa syndrome (NARP).
* Primary mitochondrial disease nuclear DNA mutations or mutations causing mtDNA destabilisation. Genetic mtDNA variants of uncertain significance, likely pathogenic, or pathogenic mutations with degrees of heteroplasmy below what can be considered to definitely cause PMD.
* General fatigue or muscle weakness due to causes other than mitochondrial disease, in the opinion of the investigator.
* Significant cardiovascular disease (e.g., sustained or symptomatic arrhythmia; dilated heart chambers or reduced function; Mobitz II atrioventricular block or greater) OR abnormal ECG that is clinically significant, as determined by the investigator. Any QTcF > 450 msec for male patients and > 470 msec for female patients is exclusionary. In the case of an exclusionary QTcF, the ECG can be repeated twice and the average of 3 QTcF intervals should be used to determine the QTcF eligibility.
* Recent history of unstable disease, inadequately controlled neurological manifestations or not recovered from stroke-like episodes including but not limited to:

  1. stroke-like episodes within the last 6 months
  2. more than 1 seizure/month within the last 6 months
  3. hospitalised for Status Epilepticus within the last 6 months
  4. more than 4 days of migraine episodes/month within the last 6 months
* History of inflammatory bowel disease, gastric erosions, peptic ulcer disease, or gastrointestinal bleeding episodes. Gastroesophageal reflux disease diagnosed by objective endoscopic or radiographic means, and clinically symptomatic at any point over the last 6 months.
* The patient has one or more clinical laboratory test values outside the reference range, based on the blood and urine samples taken at the Screening Visit, that are of potential risk to the patient's safety, or the patient has, at the Screening Visit:

  * estimated glomerular filtration rate (eGFR) calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation <30 mL/min/1.73 m2
  * a serum total bilirubin value > 1.5 times the upper limit of the reference range unless elevation is related to Gilbert's syndrome and the investigator can rule out any underlying liver dysfunction based on other tests, the patient has a Child-Pugh score ≤6, and after discussing the case with the medical monitor
  * a serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value > 2 times the upper limit of the reference range. Values between 2 and 3 times the upper limit of the reference range may be allowed if concomitant to elevation in creatine kinase as long as the investigator can rule out any underlying liver dysfunction based on other tests, the patient has a Child-Pugh score ≤6, and after discussing the case with the medical monitor
* The patient has, in the investigator's opinion, severe ataxia, neuropathy, balance problems or other medical condition that would interfere the evaluation of the 30s STS test.
* Untreated or undertreated sleep apnoea, in the opinion of the investigator.
* Use of idebenone within 14 days prior to the first dose.
* Patients have a history of unstable or severe pulmonary, immunological, oncological, hepatic disease, renal disease, or another medically significant illness other than PMD or takes medication that could, in the investigator's opinion, interfere with the assessments of safety, tolerability, or efficacy, or interfere with the conduct or interpretation of the study.
* The patient is, in the investigator's opinion, unlikely to comply with the protocol e.g. due to cognitive impairment or is unsuitable for any reason.
* The patient has an immediate family member (defined as family members residing at the same address) who participates in the study.
* Female patients with a positive pregnancy result at Screening or at Baseline.
* A patient cannot participate if they received an investigational drug 30 days or 5 half-lives prior to the Screening Visit (whichever is longer), or plans to use an investigational drug (other than the study intervention) during the study
* Hypersensitivity to the active substance or to any of the excipients or placebo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in-patient-reported fatigue symptoms and impacts on daily living measured by Patient-Reported Outcomes Measurement Information System (PROMIS®) Fatigue PMD Short Form | Baseline and 48 Weeks
  Change in t-score. Higher scores indicate greater fatigue severity.
Change in 30 Second Site-to-Stand Test. | Baseline and 48 Weeks
  Change in number of stands

SECONDARY OUTCOMES:
Change in Quality of Life in Neurological Disorders (Neuro-QoL) Lower Extremity Function (Mobility) Short Form | Baseline and 48 weeks
  Change in t-score. Higher scores indicate greater functional ability.
Change in Individual Activity Assessments - Interference | Baseline and 48 Weeks
  Assessing how much Primary Mitochondrial Disease symptoms get in the way of the ability to perform individually selected activities. A 5 point scale ranging from "No interference" to "Completely interferes"
Individual Activity Assessment - Change | 48 weeks
  Assessing the ability to perform individually selected activities compared to baseline. A 5 point scale ranging from "Much worse" to "Much better"
Change in Patient Global Impression of Severity | Baseline and 48 weeks
  Scale ranging from 1 (none) to 4 (severe).
Score on Patient Global Impression of Change | 48 weeks
  Scale ranging from 2 (much better) to -2 (much worse).
Change in Clinician Global Impression of Severity | Baseline and 48 weeks
  Scale ranging from 1 (none) to 4 (severe).
Score on Clinician Global Impression of Change | 48 weeks
  Scale ranging from 2 (much better) to -2 (much worse).
Change in Newcastle Mitochondrial Disease Adult Scale (NMDAS) - subscales I-III | Baseline and 48 weeks
  Measured on a 6-point rating scale from 0 to 5. Total score across all 3 subscales ranges from 0 to 140. Higher scores indicate more extensive and severe system involvements.
Change from baseline in Glycated haemoglobin (HbA1c) for subjects with diabetes | Baseline and 48 weeks
  mmol/mol

CONTACTS AND LOCATIONS:
Overall Officials: Amel Karaa, MD, Principal Investigator — Massachusetts General Hospital; Grainne Gorman, MD, PhD, Principal Investigator — Wellcome Centre for Mitochondrial Research, Newcastle University
Locations (23):
- United States (2):
  - Akron Children's Hospital, Akron, Ohio
  - The University of Texas Health Science Center at Houston, Houston, Texas
- Belgium (3):
  - Hopital Universitaire de Bruxelles (H.U.B)/ Academisch Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven Gasthuisberg Campus, Leuven
- Copenhagen Neuromuscular Center, Rigshospitalet, Copenhagen, Denmark
- France (5):
  - Centre Hospitalier Universitaire (CHU) de Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - Hopital Roger Salengro, CHRU de Lille, Lille
  - Centre Hospitalier Universitaire de Nice, Hopital Pasteur 2, Nice
  - CHU de NICE - Hôpital Archet 2, Nice
  - Groupe Hospitalier Pitie-Salpetriere, Paris
- Italy (5):
  - IRCCS Institute of Neurological Sciences of Bologna- Universita di Bologna, Bologna
  - Azienda Ospedaliera Universitaria Gaetano Martino Messina, Messina
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Roma
- Spain (4):
  - CIBERER- IDIBAPS, Faculty of Medicine, University of Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario de Catalunya, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (3):
  - Department of Clinical Neurosciences, Addenbrooke's Hospital, Cambridge
  - University College London Hospitals Nhs Foundation Trust, London
  - Royal Victoria Infirmary - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: Undecided